CLINICAL TRIAL: NCT06445556
Title: Uplifting Equitable Park Use and Promoting Physical Activity Among African American Families in Minnesota: A Culturally-Responsive, Community-Engaged Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MED-2024-32932
Record Dates: First submitted 2024-05-20; First posted 2024-06-06 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: This pilot study is a two-arm, parallel randomized controlled trial. 12-16 parent-child dyads will be recruited
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NatureUplift (Active Comparator): Parent-child dyads randomized to NatureUplift group
  Interventions: Behavioral: NatureUplift
- NatureUplift+Active (Experimental): Parent-child dyads randomized to NatureUplift+Active group
  Interventions: Behavioral: NatureUplift+Active

INTERVENTIONS:
Behavioral: NatureUplift — a culturally tailored, nature-based program offered at the TRPD. treatment condition will have a duration of 12 weeks, with 60 min/week of nature-based, light-intensity activities (e.g., forest bathing). Following week 12, participant dyads who were randomized to the NatureUplift intervention (i.e., delayed intervention arm) will receive access to 4 additional weeks of the NatureUplift+Active intervention.
  Arms: NatureUplift
Behavioral: NatureUplift+Active — NatureUplift plus a supplementary walking/hiking educational component. treatment condition will have a duration of 12 weeks, with 60 min/week of nature-based, light-intensity activities (e.g., forest bathing) prescribed during the NatureUplift condition and an additional 60 min/week of supplementary moderate- intensity activities (e.g., walking and hiking) prescribed during the NatureUplift+Active condition. Those who were randomized to the NatureUplift+Active intervention will continue to receive access to 4 additional weeks of the NatureUplift+Active intervention.
  Arms: NatureUplift+Active

SUMMARY:
Social injustices, such as the absence of racial representation and culturally tailored programs in parks, may further discourage African American families from accessing and using these spaces. 10 Studies are needed to investigate how exposure to more equitable greenspace environments may support physical activity (PA) among African American families. Justice-focused, park-based PA interventions hold high promise for reducing health disparities and future cardiovascular diseases (CVD) and related chronic conditions (RCC) risk, thus carrying significant implications for the fields of public health, family medicine, and urban planning.

This pilot study is a two-arm, parallel randomized controlled trial that will be conducted in partnership with community stakeholders from the Three River Park District (TRPD); TRPD parks are located in the Twin Cities region of Minnesota. This trial aims to evaluate the changes in PA, psychological health, sleep, and blood pressure among a cohort of African American parent-child dyads who will be randomized to two intervention conditions. The intervention conditions are: (1) a culturally tailored, nature-based program offered at the TRPD (hereafter, "NatureUplift"), and (2) NatureUplift plus a supplementary walking/hiking educational component (hereafter, "NatureUplift+Active"). Participant dyads will be randomized to NatureUplift or NatureUplift+Active.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for adult parents/caregivers are:

* Able and willing to provide informed consent for child
* Are the child's primary caregiver, i.e., they are the adult who spends the largest proportion of time caring for the child (e.g., cleaning, feeding, etc.) or they spent an exactly equal proportion to another caregiver (e.g., parents each with 50% of childcare responsibilities)
* Are able to read and speak English
* Self-reported Black/African American
* Live in the Twin Cities area
* Participating in less than 60 min/day and 150 min/week of PA, assessed via a modified a Godin-Shephard Leisure Time Physical Activity Questionnaire
* No contraindications to engaging in PA, assessed via the Physical Activity Readiness Questionnaire (PAR-Q+)
* Parents need to own a smartphone or a tablet to synchronize both their Fitbit and their children's Fitbit with the Fitbit application.

Inclusion criteria for youth are:

* Able and willing to provide informed assent and to comply with study requirements
* Child aged 8-12 years
* Live with the consenting parent/caregiver at least 50% of the time
* Are able to read and speak English

Exclusion Criteria:

Exclusion criteria for adult parents/caregivers are:

* Currently engaged in ≥150 min/week of PA.
* Individuals with contraindications to exercise participation as indicated by the PAR-Q+.
* A self-reported physical/mental disability that would prevent them from being able to adhere to the intervention.
* Currently pregnant or planning to become pregnant during the study period.
* Currently breastfeeding.
* Unwilling to be randomized to a study group.

Exclusion criteria for youth are:

* Currently engaged in >60 min of MVPA per day
* Individuals with contraindications to exercise participation as indicated by the PAR-Q+.
* Evidence of significant cognitive deficits or a severe, persistent psychiatric disorder (self-reported by the caregiver) that may interfere with comprehension of survey and adhere to the intervention.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-12-14 (Actual); Study Completion 2024-12-14 (Actual)

PRIMARY OUTCOMES:
Pre-/post-intervention changes in physical activity (PA) | 12 weeks
  ActiGraph GT9X will be used to measure primary outcomes (time spent in light- (LPA), moderate- (MPA), and vigorous-intensity (VPA)) Fitbits are also used, but mostly to monitor compliance and not necessarily to report on the outcome.

SECONDARY OUTCOMES:
Pre-/post-intervention changes in psychological health | 12 weeks
  assessed among child and adult participants using self-report measures, including survey items assessing for (1) perceived stress, (2) mood and affect, (3) anxiety symptoms, and (4) depressive symptoms.
Pre-/post-intervention changes in blood pressure | 12 weeks
  Pre/Post-intervention changes in blood pressure assessed among child and adult participants using a digital blood pressure monitor

CONTACTS AND LOCATIONS:
Overall Officials: Junia de Brito, PhD, MPH, MBA, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States